CLINICAL TRIAL: NCT00749138
Title: Fourteen Day Safety of Low-Dose Tamoxifen in Patients With Chronic Hepatitis C Who Have Failed Standard Medical Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bader, Ted, M.D. (Individual)
Responsible Party: Ted Bader, MD, Ted Bader, MD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102453081873
Record Dates: First submitted 2008-09-04; First posted 2008-09-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C, tamoxifen
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tamoxifen (Experimental): open label giving of tamoxifen
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: tamoxifen — giving drug tamoxifen
  Other Names: Nolvadex

SUMMARY:
A short 14 day phase 1 study examining 6 monotherapy doses of oral tamoxifen for safety in chronic HCV patients who have failed standard treatment of peginterferon and ribavirin.

DETAILED DESCRIPTION:
Six different dosages of tamoxifen will be given for 14 days with safety and viral loads being measured.

ELIGIBILITY:
Inclusion Criteria:

1. HCV RNA positive.
2. failed standard therapy

Exclusion Criteria:

1. Cirrhosis on biopsy
2. Severe medical or psychiatric conditions that would make the evaluation difficult
3. Tamoxifen is a pregnancy category D drug so pregnant women must be excluded.
4. Patients with coumadin cannot be used from a drug interaction.
5. Active use of alcohol or illegal substances -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
No significant changes in ALT or total bilirubin | 14 days

SECONDARY OUTCOMES:
HCV RNA reduction | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ted Bader, Principal Investigator — OUHSC
Locations (1):
- VA Hospital, Oklahoma City, Oklahoma, United States